CLINICAL TRIAL: NCT05757232
Title: Construction of an Ultrasound Profile and a Mammography Profile Corresponding to the Different Molecular Subtypes of Brest Cancer. A Retrospective Study of 203 Cases Diagnosed During the National Screening Campaign in 2015-2018 (PROFILS)
Brief Title: Construction of an Ultrasound Profile and a Mammographic Profile Corresponding to the Different Molecular Subtypes of Brest Cancer. A Retrospective Study
Acronym: PROFILS
Status: Completed | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: Etude PROFILS
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: screening campaign; molecular profile; tomosynthesis; ultrasound; mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancers cases diagnosed with tomosynthesis and ultrasound
- Brest cancers cases diagnosed with mammography and ultrasound

SUMMARY:
PROFILS is a retrospective, exploratory study on data collected in 203 breast cancer cases diagnosed during a national screening campaign from 2015 to 2018.

The aim of the study is to analyse histological, clinical and radiological data collected during the screening campaign to build an ultrasound profile and a mammographic profile corresponding to brest cancers' different molecular sub-types (Luminal A, Luminal B, HER2+, Triple negative) using the BI-RADS classification.

The study has the following objectives:

* To compare molecular profiles of breast cancers detected in a cohort of women diagnosed with tomosynthesis and ultrasound with molecular profiles of brest cancers detected in the cohort of women diagnosed with classical mammography and ultrasound
* To describe molecular profiles of cancers detected only with ultrasound,

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with a breast cancer
* Detection of a breast cancer during the screening campaign organized between june 2015 and july 2018 in the following geographic zones : Cantal, Haute Loire and Puys de Dôme

Exclusion Criteria:

* Patients who expressed their opposition to the use of their personal data

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The source data base of the study is from the Association Régionale des Dépistages Organisés des Cancers (ARDOC) 203 breast cancer cases have been selected in a cohort of 19 246 women who participated to the nationale breast cancer screening campaign
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Tumors' characterization using descriptive criteria of the BI-RADS classification | 3 years
  The primary outcome will be tumors' characterization using descriptive criteria of the BI-RADS classification within the framework of a mammography and an ultrasound, and then the research of a correlation with the molecular profile in 203 patientes diagnosed with a breast cancer

SECONDARY OUTCOMES:
Comparison of molecular profiles of breast cancers detected in the cohorte "mammography and ultrasound" with molecular profiles of breast cancers detected in the cohorte "tomosynthesis and ultrasound" | 3 years
  Chi 2 test or Fisher test for molecular profiles in both cohorts
Description of molecular profiles in breast cancers detected only with ultrasound | 3 years
  Descriptive statistics concerning the selection of cancers